CLINICAL TRIAL: NCT03943147
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled Evaluation of the Safety and Efficacy of BMS-986165 With Background Treatment in Subjects With Lupus Nephritis
Brief Title: An Investigational Study to Evaluate the Safety and Effectiveness of BMS-986165 With Background Treatment in Participants With Lupus Nephritis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM011-073; 2018-004142-42 (EudraCT Number)
Record Dates: First submitted 2019-04-29; First posted 2019-05-09 (Actual); Results first posted 2022-10-17 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-09

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis | interventions — deucravacitinib; Mycophenolic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BMS-986165 Dose 1 (Experimental): Specified Dose on Specified Days
  Interventions: Drug: BMS-986165; Drug: Mycophenolate Mofetil
- BMS-986165 Dose 2 (Experimental): Specified Dose on Specified Days
  Interventions: Drug: BMS-986165; Drug: Mycophenolate Mofetil
- Placebo for BMS-986165 (Placebo Comparator): Specified Dose on Specified Days
  Interventions: Drug: Placebo; Drug: Mycophenolate Mofetil
- Mycophenolate Mofetil (MMF) (Experimental): Specified Dose on Specified Days
  Interventions: Drug: Mycophenolate Mofetil

INTERVENTIONS:
Drug: BMS-986165 — Specified dose on specified days
  Arms: BMS-986165 Dose 1; BMS-986165 Dose 2
Drug: Placebo — Specified dose on specified days
  Arms: Placebo for BMS-986165
Drug: Mycophenolate Mofetil — Specified dose on specified days

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of BMS-986165 compared with placebo with regard to measures of kidney function in participants with lupus nephritis (LN).

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Meets the Systemic Lupus Erythematosus International Collaborating Clinics (SLICC) criteria for Systemic Lupus Erythematosus (SLE)
* Renal biopsy confirming a histologic diagnosis of active Lupus Nephritis (LN) International Scociety of Nephrology/Renal Pathology Society (ISN/RPS) Classes III, IV-S, or IV-G; or Class V
* Urine protein:creatinine ratio (UPCR) ≥1.5 mg/mg or UPCR ≥1 mg/mg assessed with a 24-hour urine specimen

Exclusion Criteria:

* Pure ISN/RPS Class V membranous LN
* Screening estimated glomerular filtration rate ≤30 mL/min/1.73 m^2
* Dialysis within 12 months before screening or plans for dialysis within 6 months after enrollment in the study
* End-stage renal disease

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2020-10-29 (Actual); Study Completion 2021-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (98):
- United States (40):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - The Nephrology Group, Fresno, California
  - The Regents of The University of California, Los Angeles, California
  - University of Colorado School of Medicine, Aurora, Colorado
  - Local Institution - 0029, Gainesville, Florida
  - Emory University, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Atlanta Nephrology Referral Center, Lawrenceville, Georgia
  - Northwestern Medical Faculty Foundation, Chicago, Illinois
  - The University of Chicago Medicine, Chicago, Illinois
  - Nephrology Associates of Northern Illinois and Indiana - Fort Wayne, Fort Wayne, Indiana
  - Johns Hopkins University, Office of Research Administration, Baltimore, Maryland
  - Renal and Transplant Associates of New England, PC, Springfield, Massachusetts
  - Brighton Center for Specialty Care, Brighton, Michigan
  - Clinical Research Consultants - Kansas City, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Institute for Rheumatic and Autoimmune Diseases, Summit, New Jersey
  - NewYork-Presbyterian Queens, Fresh Meadows, New York
  - Northwell Health Physician Partners at Great Neck, Great Neck, New York
  - Local Institution - 0039, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - East Carolina University Physicians, Greenville, North Carolina
  - Ohio State University, Wexner Medical Center, Columbus, Ohio
  - Local Institution - 0066, Oklahoma City, Oklahoma
  - Northeast Clinical Research Center, Bethlehem, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Local Institution - 0030, Charleston, South Carolina
  - Office of Ramesh C. Gupta, MD, Memphis, Tennessee
  - Nephrotex Research Group, Dallas, Texas
  - Dallas Nephrology Associates - North Office, Dallas, Texas
  - El Paso Medical Research Institute, El Paso, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Virginia Mason Medical Center, Seattle, Washington
  - University of Washington School of Medicine, Seattle, Washington
- Australia (2):
  - Liverpool Hospital, Liverpool, New South Wales
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Belgium (2):
  - Universitair Ziekenhuis Leuven, Leuven
  - Centre Hospitalier Universitaire de Liege Site Sart Tilman, Liège
- Canada (3):
  - Sheldon M. Chumir Health Center, Calgary, Alberta
  - Toronto Western Hospital, Toronto, Ontario
  - Centre Hospitalier Universitaire de Quebec Hospital Centre Hospitalier de IUniversite Laval, Québec, Quebec
- China (2):
  - Local Institution, Guangzhou, Guangdong
  - Local Institution, Xi'an, Shan3xi
- Czechia (2):
  - Vseobecna Fakultni Nemocnice v Praze, Prague
  - Revmatologicky Ustav, Prague
- Germany (3):
  - Universitaetsklinikum Essen, Essen
  - Medizinische Hochschule Hannover, Hanover
  - Universitatsmedizin der Johannes Gutenberg Universitat Mainz, Mainz
- Israel (3):
  - Local Institution, Haifa
  - Local Institution, Kfar Saba
  - Local Institution, Tel Aviv
- Italy (4):
  - Azienda SocioSanitaria Territoriale Fatebenefratelli Sacco, Milan
  - Local Institution - 0082, Milan
  - Universita degli Studi di Napoli Federico II, Napo
  - Istituto Scientifico di Pavia, Pavia
- Mexico (8):
  - Morales Vargas Centro de Investigacion, León, Guanajuato
  - Centro Integral de Reumatologia, Guadalajara, Jalisco
  - Investigacion Biomedica para el Desarrollo de Farmacos S.A. de C.V., Zapopan, Jalisco
  - Unidad de Investigacion de las Enfermedades Reumaticas, Mexico City, Mexico City
  - Local Institution - 0094, Mexico City, Mexico City
  - Servicios Hospitalarios de Mexico, Chihuahua City
  - Centro de Atencion e Investigacion Cardiovascular del Potosi, San Luis Potosí City
  - Hospital Central Doctor Ignacio Morones Prieto, San Luis Potosí City
- Netherlands (2):
  - Maastricht University Medical Centre, Maastricht
  - Erasmus Medisch Centrum, Rotterdam
- Russia (4):
  - Medical Center, Kemerovo
  - City Clinical Hospital #15 named after O.M. Filatova, Moscow
  - V.A. Nasonova Research Rheumatology Institute, Moscow
  - Local Institution - 0015, Saratov
- South Korea (6):
  - Local Institution, Busan
  - Local Institution - 0071, Daejeon
  - Local Institution - 0090, Gwangju
  - Local Institution - 0056, Seoul
  - Local Institution, Seoul
  - Local Institution, Suwon
- Spain (6):
  - Fundacio Puigvert, Barcelona
  - Hospital Universitari Vall dHebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Regional Universitario de Malaga Hospital General, Málaga
  - Hospital Universitario Nuestra Senora de Valme, Seville
- Taiwan (5):
  - Local Institution, Hualien City
  - Local Institution, Kaohsiung City
  - Local Institution, Taichung
  - Local Institution - 0037, Tainan
  - Local Institution, Taipei
- United Kingdom (6):
  - Brighton and Sussex University Hospitals NHS Trust, Brighton
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - University Hospitals of Leicester NHS Trust, Leicester
  - Barts Health NHS Trust, London
  - Manchester University NHS Foundation Trust, Manchester
  - Epsom and Saint Helier University Hospitals NHS Trust, Surrey

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants with an inadequate renal response to MMF may be randomized to blinded study treatment BMS-986165 3 mg BID, BMS-986165 6 mg BID, or placebo BID, as add-on therapy to MMF in Part B. No participants were randomized to receive BMS-986165 3 mg BID or placebo BID due to low enrollment.
Groups:
- Open Label MMF: All study participants receive Mycophenolate Mofetil (MMF) at a dose of 1.5 to 3.0 g/day for 12 weeks.
  Participants who meet the criteria to continue in Part B but do not meet the randomization criteria may continue on open-label MMF with or without corticosteroids.
  The following suggested target doses of MMF should be reached by the time of randomization:
  * 1.5 to 2.0 g/day for participants self-described as Asian or of Asian descent
  * 3.0 g/day for participants self-described as Black, African American, or of African descent
  * 2.0 g/day for all others
- Open Label MMF + BMS-986165: After 12 weeks of treatment with Mycophenolate Mofetil (MMF) at a dose of 1.5 to 3.0 g/day in Part A, participants meeting randomization criteria for Part B receive BMS-986165 6 mg BID + continued open-label MMF with or without corticosteroids through 52 weeks. Randomized participants may continue to receive blinded study treatment for 52 additional weeks.
Period: Open-Label MMF Run-in (Part A)
Arm/Group | Open Label MMF | Open Label MMF + BMS-986165
Started | 16 | 0
Completed | 6 | 0
Not Completed | 10 | 0
Not completed — Other reasons | 4 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Non-compliance with study drug | 1 | 0
Not completed — Protocol-specified withdrawal criterion met | 1 | 0
Not completed — Study terminated by sponsor | 3 | 0
Period: Blinded Treatment (Part B)
Arm/Group | Open Label MMF | Open Label MMF + BMS-986165
Started | 5 | 1
Completed | 2 | 1
Not Completed | 3 | 0
Not completed — Study terminated by sponsor | 3 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population for Open Label MMF includes all participants that did not meet randomization criteria in Part B. Open Label MMF + BMS-986165 includes the participant that met the randomization criteria in Part B.
Groups:
- Total: Total of all reporting groups
Arm/Group | Open Label MMF | Open Label MMF + BMS-986165 | Total
Number analyzed (Participants) | 15 | 1 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 1 | 16
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 0 | 10
  Male | 5 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 6
  Not Hispanic or Latino | 9 | 0 | 9
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 5 | 1 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Experiencing Averse Events in the Blinded Treatment Period (Part B)
Description: An adverse event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study drug and that does not necessarily have a causal relationship with this treatment. Data collected from the week 12 visit in Part A will be used for baseline values in Part B.
Time Frame: From baseline up to 52 weeks after first dose in Part B
Population: All randomized participants in Part B
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label MMF + BMS-986165
Number analyzed (Participants) | 1
Participants | 1

2. Primary Outcome: The Number of Participants With Clinically Significant ECG Abnormalities in the Blinded Treatment Period (Part B)
Description: The number of participants with clinically significant abnormalities in electrocardiograms (ECGs) parameters. The following ECG parameters will be measured: HR, PR-interval, QRS-duration, QT-interval, QTc-interval. A single 12-lead ECG will be recorded after the participant has been supine for at least 5 minutes. Data collected from the week 12 visit in Part A will be used for baseline values in Part B.
Time Frame: From baseline up to 52 weeks after first dose in Part B
Population: All randomized participants in Part B
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label MMF + BMS-986165
Number analyzed (Participants) | 1
Participants | 0

3. Primary Outcome: The Percent Change in Vital Sign Measurements in the Blinded Treatment Period (Part B)
Description: The percent change from baseline in Vital sign measurements including: blood pressure, heart rate, respiratory rate, and temperature. Blood pressure and heart rate are measured after the participant has been resting quietly for at least 5 minutes. Data collected from the week 12 visit in Part A will be used for baseline values in Part B.
Time Frame: From baseline up to 52 weeks after first dose in Part B
Population: All randomized participants in Part B
Measure: Number; unit: Percent change from baseline
Arm/Group | Open Label MMF + BMS-986165
Number analyzed (Participants) | 1
Percent change from baseline
  Diastolic Blood Pressure(mmHg) | -3.45
  Systolic Blood Pressure(mmHg | 5.22
  Heart Rate(beats/min) | 16.87
  Respiratory Rate(breaths/min) | 6.25
  Temperature(C) | -1.35

4. Primary Outcome: The Number of Participants With Abnormal Laboratory Parameters of Clinical Significance in the Blinded Treatment Period (Part B)
Description: The number of participants with abnormal laboratory parameters (Chemistry, hematology, coagulation, immunohematology) that have been considered clinically significant. Clinically relevant laboratory results are determined by the investigator. Data collected from the week 12 visit in Part A will be used for baseline values in Part B.
Time Frame: From baseline up to 52 weeks after first dose in Part B
Population: All randomized participants in Part B
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label MMF + BMS-986165
Number analyzed (Participants) | 1
Participants | 0

5. Primary Outcome: Percent Change From Baseline in 24-hour Urine Protein:Creatinine Ratio (UPCR) at Week 24 in the Blinded Treatment Period (Part B)
Description: The percent change from baseline in UPCR based on 24-hour urine collections. 24-hour urine specimens measure the levels of proteins and creatinine in urine and will be used for the UPCR at baseline (week 12) and week 24.
Time Frame: Week 24
Population: All randomized participants in Part B
Measure: Number; unit: Percent change from baseline
Arm/Group | Open Label MMF + BMS-986165
Number analyzed (Participants) | 1
Percent change from baseline | -34.86

6. Secondary Outcome: The Number of Participants With Partial Renal Response (PRR) at Week 24 in the Blinded Treatment Period (Part B)
Description: The number of participants with partial renal response (PRR) defined as ≥ 50% reduction from baseline in 24-hour Urine Protein:Creatinine Ratio (UPCR). 24-hour urine specimens measure the levels of proteins and creatinine in urine and will be used for the UPCR at baseline (week 12) and week 24.
Time Frame: Week 24
Population: All randomized participants in Part B
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label MMF + BMS-986165
Number analyzed (Participants) | 1
Participants | 0

7. Secondary Outcome: The Number of Participants With Partial Renal Response (PRR) at Week 52 in the Blinded Treatment Period (Part B)
Description: The number of participants with partial renal response (PRR) defined as ≥ 50% reduction from baseline in 24-hour Urine Protein:Creatinine Ratio (UPCR). 24-hour urine specimens measure the levels of proteins and creatinine in urine and will be used for the UPCR at baseline (week 12) and week 52.
Time Frame: Week 52
Population: All randomized participants in Part B
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label MMF + BMS-986165
Number analyzed (Participants) | 1
Participants | 0

8. Secondary Outcome: The Number of Participants With Complete Renal Response (CRR) at Week 24 in the Blinded Treatment Period (Part B)
Description: The number of participants with complete renal response (CRR) defined as a 24-hour Urine Protein:Creatinine Ratio (UPCR) ≤ 0.5 mg/mg and an estimated glomerular filtration rate (eGFR) (using the MDRD equation) ≥ 60 mL/min or ≤ 20% decrease from baseline.
Time Frame: Week 24
Population: All randomized participants in Part B
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label MMF + BMS-986165
Number analyzed (Participants) | 1
Participants | 0

9. Secondary Outcome: The Number of Participants With Complete Renal Response (CRR) at Week 52 in the Blinded Treatment Period (Part B)
Description: as for outcome 8
Time Frame: Week 52
Population: All randomized participants in Part B
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label MMF + BMS-986165
Number analyzed (Participants) | 1
Participants | 0

10. Secondary Outcome: The Number of Participants With Complete Renal Response (CRR) Plus Successful Corticosteroid Taper to ≤ 7.5 mg/Day at Week 24 in the Blinded Treatment Period (Part B)
Description: The number of participants with complete renal response (CRR) defined as a 24-hour Urine Protein:Creatinine Ratio (UPCR) ≤ 0.5 mg/mg and an estimated glomerular filtration rate (eGFR) (using the MDRD equation) ≥ 60 mL/min or ≤ 20% decrease from baseline who was also able to successfully taper corticosteroid use to ≤ 7.5 mg/day.
Time Frame: Week 24
Population: All randomized participants in Part B
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label MMF + BMS-986165
Number analyzed (Participants) | 1
Participants | 0

11. Secondary Outcome: The Number of Participants With Complete Renal Response (CRR) Plus Successful Corticosteroid Taper to ≤ 7.5 mg/Day at Week 52 in the Blinded Treatment Period (Part B)
Description: as for outcome 10
Time Frame: Week 52
Population: All randomized participants in Part B
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label MMF + BMS-986165
Number analyzed (Participants) | 1
Participants | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed from first dose to study completion (up to approximately 26 months). SAEs and Other AEs were assessed from first dose to 30 days following last dose (up to approximately 16 months)
Arm/Group | Open Label MMF | Open Label MMF + BMS-986165
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/16 | 1/1
Other Adverse Events (participants affected / at risk) | 7/16 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open Label MMF (N=16) | Open Label MMF + BMS-986165 (N=1)
COVID-19 pneumonia (Infections and infestations) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open Label MMF (N=16) | Open Label MMF + BMS-986165 (N=1)
Deafness neurosensory (Ear and labyrinth disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Gallbladder polyp (Hepatobiliary disorders) | 1 | 0
COVID-19 (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1
Blood pressure increased (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 0 | 1
Prothrombin time prolonged (Investigations) | 0 | 1
Weight increased (Investigations) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Due to low enrollment, the Sponsor chose to terminate the study on 01-Jul-2021 and consequently there is limited data available from a single randomized participant. Due to lack of sufficient data, no formal statistical analyses of endpoints were conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-06): https://cdn.clinicaltrials.gov/large-docs/47/NCT03943147/Prot_SAP_000.pdf